CLINICAL TRIAL: NCT02431455
Title: The Effect of Postoperative Incentive Spirometry on Pulmonary Function and Pulmonary Complications in Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Principal Investigator, Dmitry Nepomnayshy, Assistant Professor of Surgery TUFTS Medical School, Lahey Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-019
Record Dates: First submitted 2015-04-01; First posted 2015-05-01 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Obesity, Morbid; Complications of Bariatric Procedures; Pulmonary Atelectasis; Pneumonia
Keywords: Bariatric Surgery; obesity, morbid; incentive spirometry
MeSH Terms: conditions — Obesity, Morbid; Pulmonary Atelectasis; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Incentive Spirometry (Active Comparator): Incentive spirometry 10 times per hour while awake
  Interventions: Device: Incentive spirometer
- No Incentive Spirometry (Experimental): No incentive spirometer provided
  Interventions: Device: No incentive spirometer

INTERVENTIONS:
Device: Incentive spirometer — Incentive spirometer is provided to the patient, this is the current standard of care, and is the control arm.
  Other Names: Control
  Arms: Incentive Spirometry
Device: No incentive spirometer — No incentive spirometer is provided to the patient, this is the study arm.
  Other Names: Study
  Arms: No Incentive Spirometry

SUMMARY:
This study evaluates the omission of incentive spirometry use following bariatric surgery. Half of participants will receive an incentive spirometer while the other half will not. Oxygen saturation and pulmonary complications after surgery will be measured to examine the effectiveness of incentive spirometry.

DETAILED DESCRIPTION:
Incentive spirometry is speculated to improve pulmonary function in the postoperative period, though data to support this is lacking. Patients undergoing bariatric surgery are at increased risk for pulmonary compromise as they are obese and undergoing foregut surgery.

This study aims to examine the effect of incentive spirometry after bariatric surgery by performing a prospective randomized trial. Subjects will be randomized to either receive an incentive spirometer or not. The primary outcome measure of oxygen saturation off of supplemental oxygen will be taken preoperatively and at 6,12, and 24 hours postoperatively. Secondary outcome measures include rate of pulmonary complications, and time to wean off of supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Patients medically cleared to undergo bariatric surgery per the usual screening process

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Nepomnayshy, MD, Principal Investigator — Lahey Clinic General Surgery
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States

REFERENCES:
- [Derived] Pantel H, Hwang J, Brams D, Schnelldorfer T, Nepomnayshy D. Effect of Incentive Spirometry on Postoperative Hypoxemia and Pulmonary Complications After Bariatric Surgery: A Randomized Clinical Trial. JAMA Surg. 2017 May 1;152(5):422-428. doi: 10.1001/jamasurg.2016.4981. PMID 28097332

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Incentive Spirometry | No Incentive Spirometry
Started | 112 | 112
Completed | 112 | 112
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Incentive Spirometry | No Incentive Spirometry | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (12.4) | 45.9 (11.1) | 45.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 86 | 174
  Male | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Hypoxia 6 Hours Postoperative
Description: Number of subjects with pulse oximetry reading of < 92% with subject off of supplemental oxygen for 5 minutes with head of bed at 30°, 6 hours postoperative.
Time Frame: 6 hours postoperative
Measure: Number; unit: participants
Arm/Group | Incentive Spirometry | No Incentive Spirometry
Number analyzed (Participants) | 112 | 112
participants | 13 | 11

2. Primary Outcome: Hypoxia 12 Hours Postoperative
Description: Number of subjects with pulse oximetry reading of < 92% with subject off of supplemental oxygen for 5 minutes with head of bed at 30°, 12 hours postoperative.
Time Frame: 12 hours postoperative
Measure: Number; unit: participants
Arm/Group | Incentive Spirometry | No Incentive Spirometry
Number analyzed (Participants) | 112 | 112
participants | 6 | 9

3. Primary Outcome: Hypoxia 24 Hours Postoperative
Description: Number of subjects with pulse oximetry reading of < 92% with subject off of supplemental oxygen for 5 minutes with head of bed at 30°, 24 hours postoperative.
Time Frame: 24 hours postoperative
Measure: Number; unit: participants
Arm/Group | Incentive Spirometry | No Incentive Spirometry
Number analyzed (Participants) | 112 | 112
participants | 4 | 5

4. Secondary Outcome: Postoperative Respiratory Complication
Description: atelectasis found on chest imaging, pneumonia, or re intubation
Time Frame: entire inpatient say, usually 1 to 7 days
Measure: Number; unit: participants
Arm/Group | Incentive Spirometry | No Incentive Spirometry
Number analyzed (Participants) | 112 | 112
participants | 8 | 4

ADVERSE EVENTS:
Arm/Group | Incentive Spirometry | No Incentive Spirometry
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/112
Other Adverse Events (participants affected / at risk) | 0/112 | 0/112

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes